CLINICAL TRIAL: NCT03363971
Title: Treatment of Posttraumatic Swelling and Pain With Zhi Kang Capsule: a Multicenter, Phase IV Clinical Trial
Brief Title: Treatment of Posttraumatic Swelling and Pain With Zhi Kang Capsule
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, baoguojiang, Director of Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUPH20170988
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Soft Tissue Injuries
Keywords: soft tissue, pain
MeSH Terms: conditions — Soft Tissue Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Zhi Kang Capsule, 0.3g/capsule, oral, 4 capsules at a time, 3 times a day, half an hour after dinner, warm water delivery,treatment for 6 weeks.
  Interventions: Drug: Zhi Kang Capsule
- Control group (Placebo Comparator): Simulant agent for Zhi Kang Capsule,consistent with the appearance, color, odor, and usage of the Zhi Kang capsule, so that it can not be distinguished.oral, 4 capsules at a time, 3 times a day, half an hour after dinner, warm water delivery, treatment for 6 weeks.
  Interventions: Drug: Simulant agent for Zhi Kang Capsule

INTERVENTIONS:
Drug: Zhi Kang Capsule — 0.3g/capsule, oral, 4 capsules at a time, 3 times a day, half an hour after dinner, warm water delivery; treatment for 6 weeks.
  Arms: Experimental group
Drug: Simulant agent for Zhi Kang Capsule — 0.3g/capsule,oral, 4 capsules at a time, 3 times a day, half an hour after dinner, warm water delivery; treatment for 6 weeks.
  Arms: Control group

SUMMARY:
Zhi Kang Capsule functions for hemostasis and detumescence and can be used for traumatic bleeding, uterine bleeding, hematemesis and hematochezia.This randomized controlled trial was conducted to confirm the efficacy and safety of Zhi Kang Capsule in the treatment of posttraumatic swelling and pain,and also in a wide range of applications by open clinical observation.

DETAILED DESCRIPTION:
Limb fracture is a common disease in the Department of orthopedics, surrounding soft tissue swelling is the most common phenomenon of fracture and surgical treatment.The swelling, limb discomfort and increased pain seriously affecting the treatment effect.Therefore, prevention and treatment of limb swelling and perioperative pain is the main content of the treatment of fractures.

Post traumatic swelling and pain belong to the category of blood stasis syndrome in traditional Chinese medicine.Under the guidance of traditional Chinese medicine theory, traditional Chinese medicine plays a wide range of therapeutic effects, with a syndrome of multiple characteristics, but from the syndrome to the disease diagnosis and treatment process, more and more modern evidence based on medicine support are needed.A randomized controlled trial was carried out in the phase IV clinical trial to confirm the therapeutic effect of the capsule on posttraumatic swelling and pain. Meanwhile, an open clinical trial was conducted to evaluate the safety of the capsule in a wide range of applications.

The research subjects are patients with acute limb fractures within 2 weeks.The inclusion criteria are:(1) diagnosis of limb closed acute fracture, fracture occurred within 14 days, need for surgical treatment;(2) age ranged from 18 to 80 years old, both male and female;(3) voluntarily signed the informed consent form as the subjects.Test grouping include the capsule group and the placebo group.

The research consists of two parts: (1) the core research part: The core study was a placebo-controlled, randomized, double-blind, multicenter trial designed with 400 units of sample size, including 200 patients in the Zhi Kang Capsule group and 200 in the placebo group. The aim of the core study is to evaluate the effectiveness of test drugs. (2) the expanded research part: on the basis of core research,1800 cases were further divided into the capsule group. The aim of the expanded study was to evaluate the safety of the capsule in a large sample.

Criteria for efficacy evaluation include: pain score, swelling degree, lead flow, laboratory indicators and the first healing rate of surgical incision.All the statistical tests were two-sided, and the P value was less than or equal to 0.05, which would be considered statistically significant (except for the special description). The measurement data are described by means of mean, median, standard deviation, maximum, minimum, 25% and 75% quantiles; enumeration data or rank data are expressed in frequency and frequency.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of limb closed acute fracture, fracture occurred within 14 days, need for surgical treatment;
* age ranged from 18 to 80 years old, both male and female;
* voluntarily signed the informed consent form as the subjects.

Exclusion Criteria:

* open fracture
* multiple fractures (more than 1) or with vascular, nerve and visceral injuries
* severe primary diseases associated with heart, brain, liver, kidney, lung and hematopoietic system
* allergic constitution, mental patients
* patients with severe gastrointestinal diseases, such as ulcers; patients with severe metabolic diseases
* patients with history of alcohol addiction or drug abuse
* patients with poor compliance
* lactating women, women of pregnancy or childbearing age or male patients, do not agree to adopt effective contraceptive measures during the study period
* participants who participated in other clinical trials within the first three months of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-03-13 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 14 days
  assess the pain scores with the numerical rating scale (NRS)

SECONDARY OUTCOMES:
Swelling | 14 days
  assess the swelling degree

CONTACTS AND LOCATIONS:
Overall Officials: People's Hospital Peking University, Study Director — Peking University
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No